CLINICAL TRIAL: NCT02491346
Title: A Randomized Controlled Trial Comparing SGC and Conventional Empiric Treatment for Glucose Control in Critically Ill Patients With Mechanical Ventilation in ICU
Brief Title: A Trial Comparing SGC and Conventional Empiric Treatment for Glucose Control in Critically Ill Patients With Mechanical Ventilation in ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICU_2014-11
Record Dates: First submitted 2015-05-18; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-05

CONDITIONS: Hyperglycemia; Respiratory Failure; Critical Illness
MeSH Terms: conditions — Hyperglycemia; Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional empirical glycemic control (Active Comparator): the patients' blood glucose is controlled by physician according to their experience through insulin subcutaneous injection or insulin continuous infusion whose dosage is determinated by the physician.
  Interventions: Procedure: conventional empirical glycemic control
- SGC directed glycemic control (Experimental): the patients' blood glucose is controlled by SGC system through insulin continuous infusion whose dosage is determinated by SGC.
  Interventions: Procedure: SGC directed glycemic control

INTERVENTIONS:
Procedure: conventional empirical glycemic control — the patients' blood glucose is controlled by physician according to their experience through insulin subcutaneous injection or insulin continuous infusion whose dosage is determinated by the physician.
  Other Names: comparator group
  Arms: conventional empirical glycemic control
Procedure: SGC directed glycemic control — the patients' blood glucose is controlled by SGC system through insulin continuous infusion whose dosage is determinated by SGC.
  Other Names: SGC group
  Arms: SGC directed glycemic control

SUMMARY:
Poor glycemic control in critically ill patients can increase their mortality, while safe and efficient glucose control is laborious and time-consuming. The Space GlucoseControl which is installed with eMPC(enhanced Model Predictive Control) can get the blood glucose target range safely and effectively through regulating insulin dose rate. This study is a random controlled trial involving the patients with mechanical ventilation in intensive care unit in order to evaluate the difference of safety and efficacy of blood glucose control between SGC directed and conventional treatment. At last, the trial results can determine whether the Space GlucoseControl can control blood glucose safely and effectively in the patients with mechanical ventilation in intensive care units.

DETAILED DESCRIPTION:
Design: The study was conducted as a single-centre, open randomized controlled, parallel trial.

Study population: Adult medical ICU patients who were mechanically ventilated and assumed to require at least 3 days of intensive care were recruited. Patients fulfilling the inclusion criterion of glucose≥9.0 mM were randomly assigned using serially numbered to either the intervention group (BG control by SGC) or the control group (conventional empiric BG management). The both group aim to establish the BG levels 5.8-8.9mM.

Study protocol: BG measurements were performed using glucometer to test the fingertip capillary blood sample for the BG levels. As for patients with shock or required vasopressor, arterial BG was sampled to measure through the glucometer. Insulin [40 IU of Actrapid HM (Wanbang Biopharmaceuticals, Jiangsu province, China)/40ml of 0.9% sodium chloride] was infused intravenously applying the standard perfusor of the ICU (Perfusor®Space, B. Braun Melsungen AG, Melsungen, Germany). All trial-related activities were carried out until the end of the patient's ICU stay, or for a period of 72 hours. Meanwhile, enteral and parenteral nutrition was administrated to patients according to their condition.

Statistical analysis was performed on an intention-to-treat basis. The percentage of values in the target range (5.8-8.9mM) was defined as primary end point for the assessment of glucose control. Data are reported as mean±SD values if not otherwise indicated. Data analysis was performed using SPSS19.0.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the ICU
2. At least one BG measurement 9.0mmol/L or higher
3. Expected to stay in ICU ≥3 days;
4. Mechanical ventilation

Exclusion Criteria:

1. Aged < 18 years;
2. Admitted because of diabetic ketoacidosis or nonketotic hyperosmolar state
3. Pregnant
4. In a state in which death was perceived as imminent
5. Without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
the percentage of time within the predefined glucose the target range(5.8-8.9mmol /l) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Dr, Principal Investigator — MICU of Peking Union Medical College Hospital
Locations (1):
- MICU of Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu B, Jiang W, Wang CY, Weng L, Hu XY, Peng JM, Du B. Comparison of Space Glucose Control and Routine Glucose Management Protocol for Glycemic Control in Critically Ill Patients: A Prospective, Randomized Clinical Study. Chin Med J (Engl). 2017 Sep 5;130(17):2041-2049. doi: 10.4103/0366-6999.213422. PMID 28836546